CLINICAL TRIAL: NCT06939517
Title: Antiemetic Effect of Acupressure Wristbands for GLP-1RA Related Nausea
Brief Title: Acupressure Wristbands for GLP-1RA Related Nausea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florencia Ziemke (Other)
Responsible Party: Sponsor-Investigator, Florencia Ziemke, Founder, Medical Director, Evexia Medical
Organization: Evexia Medical (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU25020070_evexiamed
Record Dates: First submitted 2025-04-04; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Nausea
Keywords: nausea relief; acupressure wristbands; glp-1 medication; obesity
MeSH Terms: conditions — Nausea; Obesity

STUDY DESIGN:
Intervention Model Description: prospective interventional study of four weeks duration evaluating the antiemetic effect of wristbands for nausea related to GLP-1RA medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Acupressure wristband (Experimental): Study arm using acupressure wristband for nausea relief associated to GLP-1
  Interventions: Device: SeaBand

INTERVENTIONS:
Device: SeaBand — Drug-free, reusable Acupressure elastic wristbands applied to bilateral wrists for nausea relief

SUMMARY:
Nausea is a common side effect of GLP-1RA medications used for treatment of Type 2 diabetes mellitus and obesity. Current recommendations for nausea relief include the use of dietary changes and prescription anti-emetics. Acupressure wristbands Sea-Band are FDA cleared for nausea relief in other indications such as motion sickness, morning sickness in pregnancy, post-operative nausea, chemotherapy associated nausea. We hypothesized that acupressure wristbands could alleviate nausea in persons taking GLP-1RA.

DETAILED DESCRIPTION:
Nausea is the most commonly reported side effect of the class of drugs collectively known as glucagon like peptide-1 receptor agonists (GLP-1RA). GLP-1RAs are FDA approved to treat Type 2 diabetes mellitus (T2DM) and Obesity. Sea-Band is an FDA-cleared set of drug-free elastic wristbands used for nausea relief in several indications including motion sickness, morning sickness in pregnancy, post-operative nausea, chemotherapy associated nausea in persons ages 3 years old and up. The elastic wristbands have a plastic skin facing knob that apples pressure to an acupressure point called pericardium 6 (P6) located below the crease of the wrist. We hypothesize that Sea-Band can alleviate nausea in persons taking GLP-1RA. Participants on GLP-1RA medication with nausea were offered a set of Acupressure wristbands, and followed for four weeks. Weekly touch points assessed the response to nausea relief of the bands. Eligibility for the study included Adults taking GLP-1RA experiencing nausea.

ELIGIBILITY:
Inclusion Criteria:

* Adults taking GLp-1RA with nausea

Exclusion Criteria:

* Adults on GLP-1RA without nausea
* Uncontrolled GERD
* Hx of Gastroparesis
* Other nausea related conditions such as vertigo
* History of chronic use of antiemetic medication for other reasons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-04-13 (Estimated)

PRIMARY OUTCOMES:
Nausea relief | Nausea relief with use of wristbands for every recorded episode, reviewed weekly, for a total of four weeks
  Participants will be asked to apply the wristbands at the onset of nausea, and record each nausea episode using a tracker. Weekly touch points with the study team will review their number of nausea episodes, and if nausea relief was obtained.

SECONDARY OUTCOMES:
Time to onset of relief | Time to nausea relief with use of wristbands for every recorded episode, reviewed weekly, for a total of four weeks
  Participants will be asked to apply the wristbands at the onset of nausea, and record each nausea episode, confirm use of wristbands, and if time to relief was under five minutes using a tracker. Weekly touch points with the study team will review their nausea episodes. If relief was obtained, time to relief will be assessed as under or over five minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Evexia Medical, Jupiter, Florida, United States

IPD SHARING:
Plan to Share IPD: No